CLINICAL TRIAL: NCT02410603
Title: Isolating and Testing Circulating Tumor DNA and Soluble Immune Markers During the Course of Treatment for Lung Cancer
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Aaron S. Mansfield, M.D., PI, Mayo Clinic
Other Study IDs: 15-000373
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Lung Cancer; Lung Neoplasms; Cancer of Lung; Cancer of the Lung; Neoplasms, Lung; Neoplasms, Pulmonary; Pulmonary Cancer; Pulmonary Neoplasms; Carcinoma, Non-small-cell Lung; Adenocarcinoma; Squamous Cell Carcinoma
Keywords: Chemotherapy
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to explore the detection of circulating tumor DNA, soluble immune markers, and the evaluation of peripheral blood mononuclear cells (PBMC).

DETAILED DESCRIPTION:
Our plan is to collect blood from patients with advanced stage lung cancer who are scheduled to undergo systemic therapy. In this study we will utilize a novel technology for circulating tumor DNA detection in order to evaluate their presence in patients with lung cancer by comparing blood samples at six time points. We will obtain baseline blood and then collect blood at five time points during the course of the patient's chemotherapy treatments and at the end of treatment. These same blood collections will be used for the detection of soluble immune markers and evaluation of PBMCs.

ELIGIBILITY:
Inclusion Criteria:

* Advanced (non-resectable) malignancy in the thorax
* Age >18 years old
* Willing and able to provide consent
* No prior history of neoadjuvant therapy

Exclusion Criteria:

* Age <18 years old
* Unable to provide consent
* Patients with hemoglobin less than 10 g/dL (to minimize the impact of potential iatrogenic anemia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced stage cancer in the thorax who are scheduled to undergo systemic therapy at the Mayo Clinic in Rochester, MN.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2016-12; Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
The primary end point is the number and type of mutations detectable in the circulating tumor DNA blood samples. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Mansfield, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials